CLINICAL TRIAL: NCT05120973
Title: MultiSPectral fLuorescence Imaging as a Tool to Separate Healthy and Disease Related Lymphatic Anatomies During Lymph Node Dissections in Prostate Cancer.
Brief Title: Multispectral Fluorescence as a Tool to Separate Healthy and Disease Related Lymphatic Anatomies in Prostate Cancer.
Acronym: SPLIT
Status: Completed | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: N21SPL
Record Dates: First submitted 2021-11-03; First posted 2021-11-16 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Fluorescence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: Tc-ICG in the prostate (SN procedure) and fluorescein unlilateral in leg or abdominal wall
  Interventions: Procedure: multispectral imaging
- B: Free ICG bilateral in the abdominal wall
  Interventions: Procedure: fluorescence for lymphatic mapping

INTERVENTIONS:
Procedure: multispectral imaging — Sentinel node biopsy with Indocyanine Green -Technetium - Nanocolloid + fluorescein
  Groups: A
Procedure: fluorescence for lymphatic mapping — Indocyanine green injected in abdominal wall
  Groups: B

SUMMARY:
Multispectral imaging of the lymphatic draining pattern of the tumor and the abdominall wall/lower limb to evaluate technical feasibility to differentiate these patterns and in the future reduce the amount of complications that result from damage to lymphatic structures.

DETAILED DESCRIPTION:
By preventing unnecessary resection of healthy lymphatic tissue during extended lymph node dissections, the investigators will be able to reduce the degree and amount of complications that result from damage to the lymphatic structures. The investigators aim to evaluate the technical feasibility of imaging two different lymphatic drainage profiles, namely that of healthy tissue (i.e. the lower limbs/abdominal wall) and that of the primary tumour (i.e. prostate). To realize the differentiation, real-time multispectral fluorescence imaging of two spectrally different tracers (the lymphangiographic tracer fluorescein (injected in the lower limbs and abdominal wall) and sentinel node (SN) specific tracer Indocyanine Green (ICG)-99mTc-nanocolloid (injected in the tumour, followed by a control lymphoscintigraphy and SPECT/CT)) will allow for multispectral (or multicolor) fluorescence. Complementary to the routine surgical procedure, e.g. radical prostatectomy with extended pelvic lymph node dissection (ePLND), the lymphatic drainage pattern of both the tumour and of healthy tissue, i.e. lower limbs and abdominal wall, will be determined in the surgical field/surgical specimens.

ELIGIBILITY:
Inclusion Criteria Group A:

* Male, aged ≥ 18 years.
* WHO performance status 0,1, or 2.
* Written informed consent.
* Histopathologically confirmed adenocarcinoma of the prostate
* Increased risk of nodal metastases according to the Briganti 2012 nomogram (> 7%)
* Scheduled for surgical (laparoscopic) prostatectomy including ePLND-
* Suitable for RP and ePLND, as per institutional guidelines

Exclusion Criteria Group A:

* Prior abdominal or inguinal surgery (e.g. appendectomy)
* History of allergy to iodine, food or medicinal induced urticaria, asthma, eczema, or allergic rhinitis
* Hyperthyroid or thyroidal adenoma
* Kidney insufficiency
* History of oversensitivity to FLUORESCITE composites
* Patients using beta-blockers

Inclusion Criteria Group B:

* Male, aged ≥ 18 years.
* WHO performance status 0,1, or 2.
* Written informed consent.
* Histopathologically confirmed adenocarcinoma of the prostate
* Increased risk of nodal metastases according to the Briganti 2012 nomogram (> 15%)
* Scheduled for surgical (laparoscopic) prostatectomy including ePLND-
* Suitable for RP and ePLND, as per institutional guidelines

Exclusion Criteria Group B:

* Prior abdominal or inguinal surgery (e.g. appendectomy)
* History of allergy to iodine, food or medicinal induced urticaria, asthma, eczema, or allergic rhinitis
* Hyperthyroid or thyroidal adenoma
* Kidney insufficiency

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — men with prostate cancer
Study Population: Men >18 yrs with primary diagnosed prostate cancer eligible for robot assisted radical prostatectomy and lymph node dissection
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Feasibility of this intraoperative visualisation technique | During surgery
  The ability to visually differentiate the draining lymphatics of the lower limbs and abdominal wall, (LNLower limb/abdominal wall; fluorescein) from the disease associated LNs (LNprostate cancer; ICG-99mTc-nanocolloid) during lymph node dissection

SECONDARY OUTCOMES:
Anatomic localisation | During surgery
  Determine the anatomical relationship between lymphatic tumour spread and the lymphatic drainage profiles of the lower limbs and primary tumour (i.e. prostate) in relation to ePLND template.

CONTACTS AND LOCATIONS:
Overall Officials: Henk van der Poel, Prof. MD, Principal Investigator — NKI-AvL
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berrens AC, van Oosterom MN, Slof LJ, van Leeuwen FWB, van der Poel HG, Buckle T. Three-way multiplexing in prostate cancer patients - combining a bimodal sentinel node tracer with multicolor fluorescence imaging. Eur J Nucl Med Mol Imaging. 2023 Mar;50(4):1262-1263. doi: 10.1007/s00259-022-06034-x. Epub 2022 Nov 19. No abstract available. PMID 36401635